CLINICAL TRIAL: NCT05607810
Title: A Long-Term Follow-Up Study of ADVM-022 in Diabetic Macular Edema- INFINITY Extension
Brief Title: Long-Term Follow-up Study of ADVM-022 in DME (INFINITY-EXT)
Status: Active, not recruiting | Type: Observational
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADVM-022-10
Record Dates: First submitted 2022-10-21; First posted 2022-11-07 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: ADVM-022; ADVM-022-04; ADVM-022-10; AAV.7m8; Anti-VEGF therapy; Blindness; INFINITY; Gene therapy; Aflibercept (Eylea); Retinal Diseases; Eye Diseases; AAV Vector; Adverum; DME; DR; INFINITY-EXT; INFINITY-Extension; Diabetic eye disease; Long-term Extension, Long-term Follow-up, AAV vector
MeSH Terms: conditions — Diabetic Retinopathy; Blindness; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention - Subjects who received ADVM-022 in prior clinical study
  Interventions: Genetic: ADVM-022

INTERVENTIONS:
Genetic: ADVM-022 — Long term follow-up of subjects who previously received ADVM-022
  Other Names: AAV.7m8-aflibercept

SUMMARY:
This is a prospective, observational study designed to evaluate the long-term safety and tolerability of ADVM-022 in participants with diabetic macular edema (DME). Participants who previously participated in the INFINITY parent study and received a single unilateral intravitreal dose of ADVM-022 are eligible for enrollment upon completion of the end of study visit in the parent study.

DETAILED DESCRIPTION:
This is a multi-center study to evaluate the long-term safety and tolerability of a single intravitreal (IVT) injection of ADVM-022 in a preceding "parent" study, ADVM-022-04 [INFINITY]. Participants will be followed for a total of 5 years post- ADVM-022 administration (inclusive of the parent study). There is no investigational treatment administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in the ADVM-022-04 [INFINITY] (parent) study and received ADVM-022
* Must provide signed informed consent
* Must be willing and able to comply with all study procedures

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received ADVM-022 at any dose in the INFINITY study
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and non-ocular adverse events (AEs) | 168 Weeks
Severity of ocular and non-ocular AEs | 168 Weeks

SECONDARY OUTCOMES:
Time to worsening of DME disease activity | 168 Weeks
Change from Baseline in central subfield thickness (CST) and macular volume over time measured by SD-OCT | 168 Weeks
Change from Baseline in BCVA over time | 168 Weeks
Incidence of 2-step and 3-step improvement in DRSS score over time | 168 Weeks
Incidence of 2-step and 3-step worsening in DRSS score over time | 168 Weeks
Frequency of supplemental aflibercept (2mg IVT) injections over time | 168 Weeks
Occurrence of vision-threatening complications over time | 168 Weeks
Incidence of CST < 300 μm over time | 168 Weeks
Incidence of clinically significant findings via physical examinations, ocular examinations, imaging, and laboratory evaluation | 168 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adam Turpcu, Ph.D., Study Director — Adverum Biotechnologies
Locations (7):
- United States (6):
  - Adverum Clinical Site, Beverly Hills, California
  - Adverum Clinical Site, Reno, Nevada
  - Adverum Clinical Site, Philadelphia, Pennsylvania
  - Adverum Clinical Site, Austin, Texas
  - Adverum Clinical Site, Bellaire, Texas
  - Adverum Clinical Site, The Woodlands, Texas
- Adverum Clinical Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided